CLINICAL TRIAL: NCT05396365
Title: Normative Hand Grip Strength in Healthy Adult Chilean Population: Determining Labour and Anthropometric Factors.
Brief Title: Hand Grip Strength in Chilean Adults
Status: Completed | Type: Observational
Sponsor: Maria Jesus Mena-Iturriaga (Other)
Responsible Party: Sponsor-Investigator, Maria Jesus Mena-Iturriaga, Msc, Universidad del Desarrollo
Organization: Universidad del Desarrollo (Other)
Other Study IDs: Universidad del Desarrollo
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Hand Grasp
Keywords: hand grip strength; anthropometry; grip; normative values

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Dynamometry — Hand grip dynamometer measure of strength and anthropometric measurements

SUMMARY:
Context Hand grip strength (HGS) is an important parameter to assess hand function during the rehabilitation of hand injuries. HGS serves as a clinical predictor of complications after surgery.

Purpose Establish HGS reference values in healthy adult Chilean population.

Study design analytical cross-sectional.

Method 311 healthy women and men, ages 18 to 65 years participated in the study. HGS was measured with a dynamometer, according to the American Society of Hand Therapists protocol. Additionally, anthropometric and labour characteristics were registered. Kruskal-Wallis test, Wilcoxon-Mann-Whitney test and multiple linear regression were used for data analysis. Significance was set at .05.

Results Median HGS in women was 26 kg and 43 kg for men. Men demonstrated 3% more HGS on the dominant versus non-dominant hand. Women's median HGS was no different between dominant versus non-dominant hand. In men and women, manual labour activity was associated with a higher HGS. The relationships between subject anthropometric measurements and HGS were different in women versus men.

Conclusions This study determined HGS in Chilean healthy adults. Results can be used as a reference standard for clinical measures related to illness, injury and rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged between 18 and 65 years;
2. capable of adopting a seated assessment posture -

Exclusion Criteria:

1. current hand or upper limb pain;
2. history of surgery, fracture, or any condition in the upper limb that could alter hand grip strength

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy adult Chilean subjects with age between 18-65yo
Sampling Method: Probability Sample
Enrollment: 311 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Hand Grip Strength normative values | 3 months
  The subject was seated on a chair with a vertical backrest, both feet fully supported on the ground, shoulders in neutral position, arms next to the trunk, test-side elbow at 90 degrees flexion, forearm in neutral position, and wrist at 0-30 degrees dorsiflexion and 0-15 degrees ulnar deviation. The second position of the dynamometer was used for the measurement, as recommended by the ASHT. For HGS measurement, the dynamometer was positioned vertically and aligned with the forearm to maintain the forearm and wrist position as previously described

SECONDARY OUTCOMES:
Accompanying determinant factors of hand grip strength | 10 minutes
  correlate hadn grip strength with weight, height and anthropometric characteristics measurements

CONTACTS AND LOCATIONS:
Overall Officials: Phil Sizer, Phd, Study Director — Texas Tech University Health Sciences Center
Locations (1):
- Universidad del Desarrollo, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No
We don´t share Individual Participant data

REFERENCES:
- [Result] Massy-Westropp NM, Gill TK, Taylor AW, Bohannon RW, Hill CL. Hand Grip Strength: age and gender stratified normative data in a population-based study. BMC Res Notes. 2011 Apr 14;4:127. doi: 10.1186/1756-0500-4-127. PMID 21492469
- [Result] Massy-Westropp N, Rankin W, Ahern M, Krishnan J, Hearn TC. Measuring grip strength in normal adults: reference ranges and a comparison of electronic and hydraulic instruments. J Hand Surg Am. 2004 May;29(3):514-9. doi: 10.1016/j.jhsa.2004.01.012. PMID 15140498